Parent Survey Informed Consent Form NCT04152603 Approved May 19, 2022

## [Survey Tool (to be shown on the first page; survey questions will begin on the second page)]

# **BRIEF. Family Survey**

## **BRIEF: Better Research Interactions for Every Family**

# A survey research study from the University of Washington and Seattle Children's Research Institute

We are doing a survey of people who were asked if they wanted their baby to join the DIVI (Darbe plus IV Iron) research study. The survey will ask you about your thoughts and experiences being asked about the DIVI study. This survey should take about 10 minutes.

The goal of this survey is to improve how we ask people to join research. There is no benefit to you, but your responses will help us improve the process for families in the future.

At the end of the survey, you will be asked if you want to share your contact information with us so we can send you a \$25 gift card as a thank you.

You can take this survey if you were asked if your infant could join the DIVI study, **whether or not you decided to join**.

This survey is voluntary and will not affect your or your infant's care. You can stop the survey at any time. You do not have to answer any survey question if you do not wish to. The questions in this survey may remind you of a stressful time or may make you uncomfortable. If you are upset by any questions or feel you have been harmed by participating in this research, please contact us using the information below. While we will do our best to keep your information confidential, it is possible that someone outside the study team might find out that you participated in this research or see your responses.

We will remove any information that could identify you before sharing any results of this survey.

### CONFIDENTIALITY OF RESEARCH INFORMATION

We will keep your information confidential. However, if we learn that you intend to harm yourself or others, we must report that to the authorities. We will save audio recordings on secure, password-protected computers. We will remove information that could identify you before we share any results of the study.

A description of this clinical trial will be available on <a href="http://www.clinicaltrials.gov">http://www.clinicaltrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

We have a Certificate of Confidentiality from the federal National Institutes of Health. This helps us protect your privacy. The Certificate means that we do not have to give out information, documents, or samples that could identify you even if we are asked to by a court of law. We will use the Certificate to resist any demands for identifying information.

We can't use the Certificate to withhold your research information if you give your written consent to give it to an insurer, employer, or other person. Also, you or a member of your family can share information about yourself or your part in this research if you wish.

There are some limits to this protection. We will voluntarily provide the information to:

- a member of the federal government who needs it in order to audit or evaluate the research
- individuals at the institution(s) conducting the research, the funding agency, and other
  groups involved in the research, if they need the information to make sure the research
  is being done correctly;
- the federal Food and Drug Administration (FDA), if required by the FDA;
- individuals who want to conduct secondary research if allowed by federal regulations and according to your consent for future research use as described in this form;
- authorities, if we learn of child abuse, elder abuse, or the intent to harm yourself or others.

The Certificate expires when the NIH funding for this study ends. Currently this is 02/28/2026. Any data collected after expiration is not protected as described above. Data collected prior to expiration will continue to be protected.

### USING YOUR INFORMATION IN FUTURE RESEARCH

The information you share with us for this study might be used in future research. We may remove anything that might identify you from the information. If we do, that information may be used for future research without getting additional permission from you. It is also possible that in the future we may want to use or share study information that might identify you. If we do, a review board will decide whether or not we need to get additional information from you.

Questions or comments? You may contact [contact information omitted].

**Questions about your rights as a research participant?** You may contact the University of Washington Institutional Review board at hsdinfo@uw.edu or 206-543-0098.

| Please check this box to indicate you understand that this is a voluntary survey. $\Box$ | |
|---|---|
| What is your DIVI ID number? | Reference ID written into the form inviting you to take this survey |
| Click "Next Page" to go to the s | urvey. |

Version 11.00